CLINICAL TRIAL: NCT03754738
Title: Efficacy and Safety of Balloon Guide Catheter in Mechanical Thrombectomy Patients
Acronym: ESCAPE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-ESCAPE
Record Dates: First submitted 2018-11-24; First posted 2018-11-27 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Mechanical Thrombectomy; Stroke; Balloon Guide Catheter
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon guide catheter group (Experimental): mechanical thrombectomy with a balloon guide catheter group
  Interventions: Device: Balloon guide catheter
- Non-balloon guide catheter group (Active Comparator): mechanical thrombectomy with a non-balloon guide catheter group
  Interventions: Device: Non-balloon guide catheter

INTERVENTIONS:
Device: Balloon guide catheter — Use a balloon guide catheter in the mechanical thrombectomy
  Arms: Balloon guide catheter group
Device: Non-balloon guide catheter — Use a non-balloon guide catheter in the mechanical thrombectomy
  Arms: Non-balloon guide catheter group

SUMMARY:
With mechanical thrombectomy now representing standard of care for treatment of acute ischemic stroke secondary to large vessel occlusion, identifying adjunctive techniques that result in improved outcomes for patients with LVO has become an issue of increasing importance. A number of retrospective studies have demonstrated that flow arrest during the clot retrieval process results in less clot fragmentation, lower rates of distal emboli, higher revascularization rates and improved rates of good neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* A clinical diagnosis of acute stroke, with a deficit on the NIHSS of 2 points or more.
* Intracranial arterial occlusion of the distal intracranial carotid artery or middle (M1/M2) or anterior (A1/A2) cerebral artery, demonstrated with CTA, MRA, or DSA.
* Treatment can be initiated (groin puncture) within 6 hours of symptom onset.
* Planning to mechanical thrombectomy with a stenting retriever.
* Signed informed consent prior to entering study.

Exclusion Criteria:

* Moderate stenosis, severe stenosis, or occlusion of the ipsilateral extracranial carotid artery.
* Previously deployed stents in the ipsilateral carotid artery.
* Dissections of the ipsilateral carotid artery.
* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0.
* Baseline platelet count < 50.000/µL.
* Baseline blood glucose of < 50mg/dL or >400mg/dl.
* Severe, sustained hypertension (SBP > 220 mm Hg or DBP > 110 mm Hg).
* Renal insufficiency with creatinine ≥ 3 mg/dl.
* Patients in sedation and intubated patients could not be included if baseline NIHSS is not obtained by a neurologist or emergency physician prior to sedation or intubation.
* Seizures at stroke onset which would preclude obtaining a baseline NIHSS.
* Unlikely to be available for 90 days follow-up (e.g. no fixed home address, visitor from overseas).
* Subject participating in a study involving an investigational drug or device that would impact this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2018-11-25 (Estimated); Primary Completion 2019-11-25 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Distal embolization, | After mechanical thrombectomy, usually within 3 hours

SECONDARY OUTCOMES:
Modified thrombolysis in cerebral infarction 2b/3, | After mechanical thrombectomy, usually within 3 hours
Modified thrombolysis in cerebral infarction | After mechanical thrombectomy, usually within 3 hours
Modified thrombolysis in cerebral infarction 2b/3 after the first pass | After the first pass, , usually within 3 hours
First pass recanalization rate | After the first pass, , usually within 3 hours
Number of passes | After mechanical thrombectomy, usually within 3 hours
Procedure time | From the procedure start to the end, usually within 3 hours
National Institutes of Health Stroke Scale | 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Symptomatic intracranial hemorrhage | 24 hours
Modified Rankin Scale | 90 days
  Scores on the modified Rankin scale of functional disability range from 0 (no symptoms) to 6 (death).
Mortality | 90 days

OTHER OUTCOMES:
Safety (occurrence of adverse events and serious adverse events) | 7 days

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Suzhou Municipal Hoapital, Suzhou, Anhui
  - Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Lu He hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Nanyang City Center Hospital, Nanyang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Derived] Ma H, Che R, Zhang Q, Yu W, Wu L, Zhao W, Li M, Wu D, Wu C, Ji X. The optimum anticoagulation time after endovascular thrombectomy for atrial fibrillation-related large vessel occlusion stroke: a real-world study. J Neurol. 2023 Apr;270(4):2084-2095. doi: 10.1007/s00415-022-11515-y. Epub 2023 Jan 3. PMID 36596867